CLINICAL TRIAL: NCT04000256
Title: Understanding Experiences of People With Spinal Cord Injury Undergoing Activity-based Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 19G.279
Record Dates: First submitted 2019-06-17; First posted 2019-06-27 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries; Telerehabilitation; Qualitative
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Cord Injury: The data during the first visit involves questionnaires, performance and observational measures for baseline evaluation. The 2nd to 8th visit involves feedback survey and interview data collection based on experiences of participants undergoing activity-based training using upper extremity rehabilitation equipment.
  Interventions: Behavioral: Activity based rehabilitation

INTERVENTIONS:
Behavioral: Activity based rehabilitation — Activity based rehabilitation for the upper extremity involves various gross and fine movements, reach and object transportation, and object manipulation. The rehabilitation equipment used during training will include gaming and instrumented training equipment, conventional table-top tasks, and exercise aids.

SUMMARY:
Incomplete cervical spinal cord injury (SCI) makes up half of all the newly admitted patients. For these individuals, the use of their upper limbs is critical for managing daily activities and self-care and impacts their quality of life. For home-based monitored rehabilitation, also called telerehabilitation, there are various rehabilitation equipment that are used. No studies have systematically gathered information regarding the perceptions of individuals with SCI regarding these equipment, training, and feasibility within the home. Further, their perceptions of the usability of high vs low end equipment is also not explored. In this study, investigators plan to gather survey and interview data from individuals with SCI regarding their experience with using rehabilitation equipment that uses games, muscle stimulation, and object manipulation. This study will inform the development of a tele-rehabilitation intervention in the future.

DETAILED DESCRIPTION:
Incomplete cervical spinal cord injury (SCI) makes up half of all the newly admitted patients. The overall prognosis for walking is better than the upper limb recovery in incomplete tetraplegia. Upper limb deficits result in difficulty in managing daily activities and self-care and impacts quality of life. Rehabilitation of the upper limb involves high intensity repetitive activities that are directed to a specific task. The demands of these programs can be up to 5 hours of therapy, 5 days a week for 12 weeks. Home-based therapies augmented by tele-rehabilitation presents a more realistic alternative to clinic-based application of these programs due to transportation and time commitment. However, engaging and motivating therapy options are needed for home to enhance client outcomes and improve compliance. Some of the latest equipment provides this capability and engages the patient using games for training. However, high equipment cost limits its widespread use.

In this study, we will engage individuals with cervical SCI in a 4-week (8 visit) evaluation of a variety of training protocols to gather information on their perceptions regarding motivation, engagement, and challenge it offers; its ability to address limitations they experience; and its feasibility within the home.

The long-term goal of this National Institute of Disability Independent Living and Rehabilitation (NIDILRR) funded Spinal Cord Injury Model System (SCIMS) project is to develop an engaging and evidence-informed intervention for home-based upper limb activity-based rehabilitation in individuals with spinal cord injury (SCI). A review of literature was recently conducted by the research team to get a scope of the evidence related to current activity-based therapies and the equipment used to deliver these programs. There is insufficient information about the value of high-end equipment involving games relative to lower cost alternatives, or the perceptions of clients regarding the use of various technologies related to motivation, engagement, appropriate level of difficulty and feasibility within the home. This lab-based study aims to understand the experiences related to rehabilitation training and high and low end equipment for upper limb activity-based rehabilitation in individuals with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Motor incomplete cervical SCI, neurologic levels C1-C7
2. Atleast one arm with active shoulder flexion (reach with gravity eliminated) and atleast one grasp pattern/able to move fingers
3. At least 6 months post injury
4. At least one arm with greater than 50% normal passive range of motion in all upper limb joints, excluding the interphalangeal joints of the fingers
5. Medically stable with no contraindications to the activities or to sitting
6. 18 years of age or older

Exclusion Criteria:

1. Uncontrolled pain in the upper limbs
2. Upper extremity amputations
3. Unable to commit to at least 3 visits
4. Surgical procedures (e.g., tendon transfers) or orthopedic trauma (e.g., fracture) within the past 3 months
5. Other neurological conditions
6. Mechanical Ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years or older with chronic stable cervical spinal cord injury affecting one or both arms
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
10-item questionnaire | Week 4
  Quantitative feedback using a 10-question survey regarding experiences with the rehabilitation training and equipment for feasibility, motivation, engagement and difficulty.

SECONDARY OUTCOMES:
Qualitative interview | Week 4
  Interview to explore further the experiences with rehabilitation training and equipment.
Qualitative interview | Week 2
  Interview to explore further the experiences with rehabilitation training and equipment.
10-item questionnaire | Week 2
  Quantitative feedback using a 10-question survey regarding experiences with the rehabilitation training and equipment for feasibility, motivation, engagement and difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Marino, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Chapman University, Orange, California
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Participant data from both sites will be pooled for analysis and reporting of results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: De-identified data only

REFERENCES:
- [Background] Szturm T, Peters JF, Otto C, Kapadia N, Desai A. Task-specific rehabilitation of finger-hand function using interactive computer gaming. Arch Phys Med Rehabil. 2008 Nov;89(11):2213-7. doi: 10.1016/j.apmr.2008.04.021. PMID 18996252
- [Background] Gauthier LV, Kane C, Borstad A, Strahl N, Uswatte G, Taub E, Morris D, Hall A, Arakelian M, Mark V. Video Game Rehabilitation for Outpatient Stroke (VIGoROUS): protocol for a multi-center comparative effectiveness trial of in-home gamified constraint-induced movement therapy for rehabilitation of chronic upper extremity hemiparesis. BMC Neurol. 2017 Jun 8;17(1):109. doi: 10.1186/s12883-017-0888-0. PMID 28595611
- [Background] Thielen CC, Marino RJ, Duff S, Kaplan G, Mulcahey MJ. Activity-based Rehabilitation Interventions of the Neurologically Impaired Upper Extremity: Description of a Scoping Review Protocol. Top Spinal Cord Inj Rehabil. 2018 Summer;24(3):288-294. doi: 10.1310/sci2403-288. PMID 29997431
- [Derived] Bell A, Grampurohit N, Kains G, Marino RJ. Developing guiding principles for technology-based rehabilitation program by engaging people with motor incomplete tetraplegia. J Neuroeng Rehabil. 2022 Nov 24;19(1):128. doi: 10.1186/s12984-022-01096-2. PMID 36424612